CLINICAL TRIAL: NCT05855473
Title: Effects of Auricular Acupuncture on Fatigue, Energy, and Well-Being Among Intensive Care Nurses: A Randomized Controlled Trial
Brief Title: Auricular Acupuncture on Fatigue, Energy and Well-Being in Intensive Care Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Havva SERT, Associate Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 45/08.06.2022
Record Dates: First submitted 2023-04-06; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Fatigue
Keywords: intensive care nurses; acupuncture; fatigue; well-being
MeSH Terms: conditions — Fatigue | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Semi-permanent needle (Experimental): Five sessions of unilateral auricular acupuncture were applied alternately to the right and left ears, once a week, to the intensive care nurses in the semi-permanent needle group. Semi-permanent needles placed on the acupuncture points of the nurses' ears remained for one week with adhesive tapes. In the sessions in the following weeks, semi-permanent needles were replaced with new ones. Shen men (TF4), Sympathetic (AH6a), Lung, Liver (CO12) Kidney point (CO10) were applied to five specific points in the ear in accordance with the NADA protocol.
  Interventions: Other: Auricular acupuncture
- Seed (Experimental): Five sessions of unilateral auricular acupuncture were applied alternately to the right and left ears, once a week, to the intensive care nurses in the seed group. Seeds placed on the acupuncture points of the nurses' ears remained for one week with adhesive tapes. In the sessions in the following weeks, seeds were replaced with new ones. The seed group was asked to apply pressure on the bands three times a day, 15 times each time. Shen men (TF4), Sympathetic (AH6a), Lung, Liver (CO12) Kidney point (CO10) were applied to five specific points in the ear in accordance with the NADA protocol.
  Interventions: Other: Auricular acupuncture
- Control (No Intervention): This group received no intervention.

INTERVENTIONS:
Other: Auricular acupuncture — The NADA protocol used in this study uses five specific points on the ear: Shen men, sympathetic autonomic, lung, liver, and kidney. Using this protocol, semi-permanent needles and seeds were placed unilaterally at five specific points in the ear by a specialist physician certified in acupuncture.
  Arms: Seed; Semi-permanent needle

SUMMARY:
Notably, no acupuncture intervention studies have aimed at reducing the fatigue level and increasing the energy of the nurses working in the ICU. For this reason, this study aims to investigate the effects of auricular acupuncture applied to nurses working in the ICU, who work at a critical point in patient care in our country, work with intense work tempo, experience excessive stress, tension, fatigue, and are open to psychosocial problems such as depression and burnout, on fatigue and energy levels. This study can significantly contribute to the literature on managing the physical and psychosocial issues associated with fatigue and that similar intervention programs can be expanded in working life. This study aimed to determine the effect of auricular acupuncture applied to intensive care nurses on fatigue, energy and well-being. This was a single-blind, randomized controlled clinical study. The study was conducted in three groups: semi-permanent needle acupuncture (intervention), seed acupuncture (intervention), and a control group.

DETAILED DESCRIPTION:
A stratified randomization method was used to determine intervention, placebo and control groups. It was ensured that the nurses were evenly distributed to the groups according to their age, working year and baseline fatigue scores. A computer-generated (https://www.randomizer.org/) sorting was used to allocate the groups homogeneously.

The intervention groups received five sessions of auricular acupuncture with semi-permanent needles and seeds once a week. Semi-permanent needles and seeds placed in nurses' ear acupuncture points stayed for one week. In the sessions in the following weeks, semi-permanent needles and seeds were replaced with new ones. Nurses were reminded to remove the semi-permanent needle and seed tapes 24 hours before the scheduled session. They are also instructed to remove it beforehand if there is any discomfort, itching or any sign of allergy. Placement of the semi-permanent needles and seed tapes took approximately five minutes per session. Before each session for the semi-permanent needle group, the ears of the participants were cleaned with a 70% alcohol wipe and sterile, fine-caliber, disposable semi-permanent needles were used. A similar application was made to the seed group and they were asked to apply pressure on the bands three times a day, 15 times each time.

These were placed unilaterally on five specific points in the ear (ShenMen, sympathetic, liver, kidney, lung) by a certified specialist in acupuncture using the National Acupuncture Detoxification Association (NADA) protocol. Since the body or organs have an emotional component and can be adversely affected by excessive and prolonged emotions, these ear points were chosen to facilitate the release of negative/toxic emotions from the organs. This process was thought to help the treated participant return to balance and increase energy and well-being by giving a feeling of calm instead of stress and anxiety. Shen men (TF4) and Sympathetic (AH6a) points can regulate the sympathetic and parasympathetic nervous systems to effectively reduce patient tension and anxiety. In addition, the TF4 point reduces anxiety, while the AH6a point calms excessive sympathetic activity. Both of these points help increase parasympathetic activation by balancing the sympathetic/parasympathetic branches of the autonomic nervous system. Low mood and lethargy are improved by stimulating the liver (CO12). Kidney point (CO10) is a point that has a strengthening effect by relieving mental weakness, fatigue and headaches and stimulating kidney functions. Combining these ear acupuncture points can increase the energy and blood flow of the organs, thereby relieving the patient's fatigue.

Data were collected at baseline and at the end of the intervention (week 5) using the Chalder Fatigue Scale, Subjective Vitality Scale, and Well-being Scale.

ELIGIBILITY:
Inclusion Criteria:

* Working as a nurse in the intensive care unit for at least 6 months.
* No physical disability
* Those who do not have a neurological diagnosis (having SVO, epilepsy, multiplesclerosis, etc.)
* No psychiatric diagnosis
* On the ear skin at the application site; no lesions such as infection, ulcer, irritation, rash, scar and
* Nurses who volunteered to participate in the study

Exclusion Criteria:

* Patients followed up with the diagnosis of end-stage renal disease, COPD, advanced heart failure, chronic liver disease, musculoskeletal problem, hypothyroidism and depression.
* Those who have physical and mental health problems that prevent communication
* Bleeding disorder or taking anticoagulant therapy
* pregnant
* Nurses who received any medical treatment or applied complementary methods (relaxation exercise, yoga, massage, etc.) during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Fatigue at five weeks | Baseline, 5th week (after the intervention)
  Chalder Fatigue Scale was used to evaluate the fatigue level of intensive care nurses. The scale consists of 11 items in total, including a 7-item physical fatigue subsection and a 4-item mental fatigue subsection. Participants are asked to answer the statements using a four-point Likert scale. Scoring is made between 0-3 and the total score varies between 0-33. High scores indicate greater fatigue severity.
Change from Baseline Energy Level at five weeks | Baseline, 5th week (after the intervention)
  Subjective Vitality Scale was used to evaluate the energy level of intensive care nurses. The scale, which is a 7-point Likert scale (1 strongly disagree-7 strongly agree), consists of seven items. The sum of the scores in the scale ranges from 7 to 49. High scores obtained from the scale indicate that the individual's subjective vitality level is high.
Change from Baseline Well-being at five weeks | Baseline, 5th week (after the intervention)
  Well-Being Scale was used to evaluate the well-being of intensive care nurses. Participants are expected to express their views on the scale items in a 7-point Likert-type rating ranging from 1-strongly disagree to 7-strongly agree. The highest score that can be obtained from the scale is 56, and the lowest score is 8. High scores obtained from the scale indicate that the level of well-being of the relevant individual is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No